CLINICAL TRIAL: NCT00540254
Title: Behavioral Insomnia Therapy With Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00002157; R21NR010539 (NIH); NIH: 1 R21 NR010539-01A1
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Fatigue Syndrome; Behavioral Therapy Targeted to Sleep Problems
Keywords: Chronic Fatigue; Insomnia; Cognitive Behavioral Therapy
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Cognitive Behavioral Therapy (CBT) + Insomnia plus Usual Care for Chronic Fatigue Syndrome -continues standard care for Chronic Fatigue Syndrome plus 4 sessions of CBT targeted for insomnia/sleep problems
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Arm 2 (Active Comparator): Usual Care for Chronic Fatigue Syndrome (Active Control Group) - continues standard care for Chronic Fatigue Syndrome and comes to the sleep lab for bi-weekly sessions to discuss sleep problems and to review weekly sleep logs
  Interventions: Other: Usual Care for Chronic Fatigue Syndrome (Active Control Group)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) + Insomnia plus Usual Care for Chronic Fatigue Syndrome -continues standard care for Chronic Fatigue Syndrome plus 4 sessions of CBT targeted for insomnia/sleep problems
  Arms: Arm 1
Other: Usual Care for Chronic Fatigue Syndrome (Active Control Group) — Usual Care for Chronic Fatigue Syndrome (Active Control Group) - continues standard care for Chronic Fatigue Syndrome and comes to the sleep lab for bi-weekly sessions to discuss sleep problems and to review weekly sleep logs
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine how best to manage the sleep problems of people with Chronic Fatigue Syndrome. This study is being conducted to determine how improvements in sleep affect other Chronic Fatigue symptoms including pain, fatigue, and mood as well as a person's sense of general well-being.

DETAILED DESCRIPTION:
Chronic Fatigue Syndrome (CFS) is a prevalent, debilitating, and poorly understood condition that contributes to impaired functioning and increased health care utilization. The vast majority of CFS patients complain of unrelenting sleep disturbances (e.g., sleep onset insomnia and/or sleep maintenance insomnia) that could exacerbate symptoms such as fatigue, mood disturbance, and reduced quality of life. Research with normal sleepers and insomnia sufferers has demonstrated that sleep disruption adversely affects those systems hypothesized to be important in CFS (e.g., neuroendocrine and autonomic systems). Insomnia appears to be a perpetuating factor in CFS, as insomnia appears to develop as a comorbid condition that interacts with and worsens CFS. Perhaps because the insomnia of CFS patients traditionally has been viewed as a secondary symptom rather than as a comorbid disorder, the sleep-specific treatment needs of CFS patients have been largely ignored. In fact, there have been few studies conducted to test sleep-focused therapies with CFS patients. Both our clinical observations and our preliminary studies suggest that those with CFS display sleep targets (i.e., increased time-in-bed, decreased daytime activity) that are common to those with Primary and other comorbid insomnias. These phenomena are known to perpetuate sleep problems, and likely account for the chronic insomnia among CFS patients. Given the high prevalence and cost associated with CFS, as well as its complex clinical picture, interventions that directly address perpetuating mechanisms would likely improve the sleep and general prognosis for these patients.

The proposed randomized clinical trial will allow us to test the effects of CBT for Insomnia on sleep and waking functions among CFS patients. Positive results could lead to enhanced CFS outcomes by treating the comorbid insomnia effectively.

The consent form for this study will provide participants with information about who will provide their care during the study, the purpose of the study, the number of participants expected in the study, what is required of participants in the study, information about random assignment to study groups, how long participation in the study will last, the risks associated with the study, possible benefits of participation, alternatives for treatment other than participation in this study, information about confidentiality, costs to the participants associated with the study, compensation for participation, and who to contact if there questions about the study or injuries related to the study, the right to stop participating and withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Fatigue Syndrome and Insomnia
* meet diagnostic criteria for insomnia
* be diagnosed with CFS by the Study Physician using CDC criteria
* must be in current treatment for CFS (we can provide referrals if needed).
* under medical care for a minimum of 6 weeks with a stable medication regimen for > 1 month.

Study patients can have comorbid depression (as long as it is not bipolar, melancholic or psychotic) or fibromyalgia. They can be taking sleep medications.

Exclusion Criteria:

* Those with untreated medical disorders that could account for the fatigue, or affect sleep. Medical conditions that would exclude a participant include:

  * organ failure resulting from conditions such as emphysema, cirrhosis, cardiac failure, chronic renal failure
  * chronic infections, including AIDS, and hepatitis B or C
  * rheumatic and chronic inflammatory diseases that could account for the fatigue: including systemic lupus erythematosis, Sjogren's syndrome, rheumatoid arthritis, inflammatory bowel disease, chronic pancreatitis
  * major neurologic diseases (e.g., multiple sclerosis, neuromuscular diseases, epilepsy or other diseases requiring ongoing medication that could cause fatigue, stroke, head injury with residual neurologic deficits)
  * diseases requiring systemic treatment (e.g., organ or bone marrow transplantation, systemic chemotherapy, radiation of brain, thorax, abdomen, or pelvis)
  * untreated major endocrine diseases (e.g., hypopituitarism, adrenal insufficiency)
  * being on medications with known fatigue side effects or medications that have not been stable for at least one month
  * inadequately-treated hypothyroidism
  * untreated or unstable diabetes mellitus
  * active infection
  * pregnancy, 1-3 months post-partum or breast feeding
  * within 6 months post-operation for a major surgical procedure
  * within 3 months post-operation of minor surgery
  * major infections, such as sepsis or pneumonia until 3 months post-resolution
  * major conditions whose resolution may be unclear for at least 5 years (e.g., myocardial infarction, heart failure)
  * terminal conditions
  * severe obesity as defined as a body mass index (weight in kilograms/height in meters)2 > 40
  * elective surgery planned during the trial
* We will exclude those who meet DSM-IV criteria currently or in the past 5 years for psychotic or melancholic Major Depression, bipolar disorders, schizophrenia, or eating disorders, alcohol or substance abuse or dependence (e.g., dependence on benzodiazepines or any other substance)
* We will exclude those meeting criteria for Narcolepsy, Restless Legs Syndrome, a Circadian Rhythm Disorder, or sleep apnea and/or hypopnea.
* We will exclude those with a medication change within the last month to ensure participants are on a stable dose and regimen of medication. *Once potential patients have had a stable medication regimen for > 1 month, participants can enter the trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
total wake time | Measures taken at baseline, mid-treatment, immediate post-treatment, one-month follow-up
total sleep time | Measures taken at baseline, mid-treatment, immediate post-treatment, one-month follow-up
sleep efficiency | Measures taken at baseline, mid-treatment, immediate post-treatment, one-month follow-up
beliefs about sleep | Measures taken at baseline, mid-treatment, immediate post-treatment, one-month follow-up
sleep habits | Measures taken at baseline, mid-treatment, immediate post-treatment, one-month follow-up

SECONDARY OUTCOMES:
actigraphy (measurement of activity) | Measures taken at baseline, mid-treatment, immediate post-treatment, one-month follow-up
scores on measures of fatigue, mood, anxiety, quality of life, chronic fatigue syndrome symptoms, fibromyalgia symptoms, medication usage | Measures taken at baseline, mid-treatment, immediate post-treatment, one-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, M.D., Study Director — Duke University; Mark Mayo, Principal Investigator — Duke University; Pam Smith, Principal Investigator — Duke Medical Center
Locations (1):
- Duke University Medical Center - Insomnia and Sleep Disorders Lab, Durham, North Carolina, United States

REFERENCES:
- [Background] Waters WF, Hurry MJ, Binks PG, Carney CE, Lajos LE, Fuller KH, Betz B, Johnson J, Anderson T, Tucci JM. Behavioral and hypnotic treatments for insomnia subtypes. Behav Sleep Med. 2003;1(2):81-101. doi: 10.1207/S15402010BSM0102_2. PMID 15600131
- [Background] Carney CE, Edinger JD. Identifying critical beliefs about sleep in primary insomnia. Sleep. 2006 Apr;29(4):444-53. PMID 16676777
- [Background] Edinger JD, Wohlgemuth WK, Radtke RA, Marsh GR, Quillian RE. Cognitive behavioral therapy for treatment of chronic primary insomnia: a randomized controlled trial. JAMA. 2001 Apr 11;285(14):1856-64. doi: 10.1001/jama.285.14.1856. PMID 11308399
- [Background] Edinger JD, Wohlgemuth WK, Krystal AD, Rice JR. Behavioral insomnia therapy for fibromyalgia patients: a randomized clinical trial. Arch Intern Med. 2005 Nov 28;165(21):2527-35. doi: 10.1001/archinte.165.21.2527. PMID 16314551